CLINICAL TRIAL: NCT01084954
Title: Validation of a Simple and Cost-Effective Nucleic Acid Test for HIV Detection
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: 040907
Record Dates: First submitted 2010-03-09; First posted 2010-03-11 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2015-08

CONDITIONS: HIV; HIV Infections
Keywords: HIV validation helicase-dependent amplification
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Validate a simple and cost-effective Nucleic Acid Test for HIV Detection in order to develop a rapid, highly sensitive and specific, one-stage test for the diagnosis of HIV infection. Blood samples collected will be assayed using the BioHelix Corporation helicase-dependent amplification or the Cepheid Xpert HIV-1 Quant Assay. A false negative or false positive rate of >1.0% would make this test unacceptable as a screening test for HIV viremia.

ELIGIBILITY:
Inclusion Criteria:

* Current patient in the Medical Faculty Associates Infectious Diseases (ID) clinic with known HIV infection
* Suspected to be viremic at the time of their clinic visit based on history and/or current symptoms
* Able to provide informed consent
* 18 Years or older

Exclusion Criteria:

* Patient unable to provide informed consent.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infectious Disease Clinic, HIV Positive patients
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2009-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Validation of a Simple and Cost-Effective Nucleic Acid Test for HIV Detection | Participation will last 1 hour for subjects to consent and provide a single blood sample.
  A false negative or false positive rate of > 1.0% would make this test unacceptable as a screening test for HIV viremia.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Simon, M.D., Ph.D., Principal Investigator — George Washington University
Locations (1):
- The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No